CLINICAL TRIAL: NCT00994617
Title: Monotherapy Versus Dual Therapy for Initial Treatment for Hypertension
Acronym: Pathway 1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Morris Brown, Prof Morris Brown, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-007749-29
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Essential Hypertension
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Essential Hypertension | interventions — hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy (Experimental): Patients treated with combination therapy of Hydrochlorthiazide plus Losartan. Losartan will be force-titrated from 50 to 100mg, Hydrochlorothiazide will be force-titrated from 12.5mg to 25mg
  Interventions: Drug: Losartan and hydrochlorothiazide
- Monotherapy (Active Comparator): Initial monotherapy Hydrochlorothiazide 12.5mg -25mg Crossed over with Losartan 50 -100mg at 8 weeks
  Interventions: Drug: Hydrochlorothiazide switched over with Losartan at 8 weeks

INTERVENTIONS:
Drug: Losartan and hydrochlorothiazide — Losartan 50 -100mg Hydrochlorothiazide 12.5mg -25mg
  Arms: Combination Therapy
Drug: Hydrochlorothiazide switched over with Losartan at 8 weeks — Hydrochlorothiazide 12.5-25mg crossed over with Losartan 50-100mg
  Arms: Monotherapy

SUMMARY:
To test whether the current custom of initiating treatment for hypertension with a single drug is less effective in the short-term than initial combination therapy, and results in the eventual need for comparatively more antihypertensive drug therapy.

DETAILED DESCRIPTION:
To determine if patients randomised to more aggressive (combination therapy) treatment for the initial treatment of hypertension have better blood pressure control compared to those randomised to less aggressive (monotherapy) treatment despite subsequent add-on treatment being similar in each group. This will test the hypothesis that monotherapy patients 'never catch up' with combination therapy patients.

1. To determine if this 'never catch-up' phenomenon of improved BP control persists for at least one year.
2. To understand the underlying mechanism of improved BP control; specifically:

   1. To determine if it is due to haemodynamic compensation, such as increased sodium retention and volume expansion.
   2. To determine if it is due to increased peripheral resistance.
3. To understand the predictors of BP control i.e. age, baseline renin status, sodium status and plasma volume.
4. To validate the National Institute for Clinical Excellence / British Hypertension Society joint guideline ACD algorithm by comparing BP control in the monotherapy crossover arm of phase 1 and to correlate this with age (≤ 55 or > 55y), and baseline characteristics such as renin.
5. To determine the safety and tolerability of a strategy of prescribing combination therapy as the initial step versus monotherapy as the initial step.

ELIGIBILITY:
Patients must meet ALL inclusion criteria

1. Aged 18-79
2. Male subjects or female subjects taking adequate contraception such as the oral contraceptive pill, an intra uterine device or who are surgically sterilised or postmenopausal Females
3. BP ≥150 mmHg (systolic) OR ≥ 95 mmHg (diastolic). Patients may be included if the PI anticipates BP criteria for inclusion will be met at randomisation
4. Either never-treated or received a maximum of one antihypertensive drug class in the previous year

Patients will be excluded for ANY ONE of the following reasons

1. Clinic SBP > 200 mmHg or DBP > 120 mmHg, with PI discretion to override if home BP measurements are lower
2. Secondary or accelerated phase hypertension
3. eGFR < 45 mls/min
4. Contra-indication or previous intolerance to any trial therapy
5. Failure to record required home BP readings during placebo run-in.
6. Significant co-morbidity (investigator opinion but to include alcoholism, terminal illness, documented non-attendance at clinics etc)
7. Diabetes type 1
8. Plasma K+ outside normal range on two successive measurements during screening
9. Requirement for treatment with ≥2 drugs (which can be a CCB and/or {ACEi OR ARB OR direct renin inhibitor OR β-blocker}) in order to reduce blood pressure to ≤180/120 mmHg
10. Requirement for diuretic therapy (other than for hypertension)
11. Requirement for ACE inhibitor (or ARB) therapy (other than for hypertension)
12. Absolute contra-indications to any of the study drugs (listed on their data-sheet)
13. Current therapy for cancer
14. Anticipation of change in medical status during course of trial (e.g. planned surgical intervention requiring >2 weeks convalescence , actual or planned pregnancy)
15. Inability to give informed consent
16. Participation in a clinical study involving an investigational drug or device within 4 weeks of screening.
17. Any concomitant condition that, in the opinion of the investigator, may adversely affect the safety and/or efficacy of the study drug or severely limit the subject's lifespan or ability to complete the study (eg, alcohol or drug abuse, disabling or terminal illness, mental disorders).
18. Treatment with any of the following prohibited medications:

    1. Oral corticosteroids within 3 months of screening. Treatment with systemic corticosteroids is also prohibited during study participation.

       Chronic stable or unstable use of non-steroidal anti-inflammatory drugs (NSAIDs) other than acetylsalicylic acid is prohibited. Chronic use is defined as >3 consecutive or nonconsecutive days of treatment per week. In addition, the intermittent use of NSAIDs is strongly discouraged throughout the duration of this study. If intermittent treatment is required, NSAIDs must not be used for more than a total of 2 days. For all subjects requiring analgesic or anti-pyretic agents, the use of paracetamol is recommended during study participation.
    2. The use of short-acting oral nitrates (eg, sublingual nitroglycerin) is permitted; however, subjects should not take short-acting oral nitrates within 4 hours of screening or any subsequent study visit.
    3. The use of long-acting oral nitrates (eg, Isordil) is permitted; however, the dose must be stable for at least 2 weeks prior to screening and randomisation.
    4. The use of sympathomimetic decongestants is permitted; however, not within 1 day prior to any clinic visit/BP assessment.
    5. The use of theophylline is permitted; however, the dose must be stable for at least 4 weeks prior to screening and throughout study participation.
    6. The use of phosphodiesterase (PDE) type V inhibitors is permitted; however, subjects must refrain from taking these medications within 1 day of screening or any subsequent study visit.
    7. The use of alpha-blockers is not permitted - with the exception of afluzosin and tamsulosin for prostatic symptoms

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean home systolic BP for the group treated initially with monotherapy compared to the group treated initially with combination therapy. | 1 year

SECONDARY OUTCOMES:
A comparison the proportion of patients who drop out of the trial at any stage after randomisation or who require further antihypertensive treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Professor MJ Brown, FMedSci, Principal Investigator — University of Cambridge
Locations (13):
- United Kingdom (13):
  - Professor Morris Brown, Cambridge, Cambridgeshire
  - NHS Ayrshire, Ayrshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Tayside/University of Dundee, Dundee
  - NHS Lothian/University of Edinburgh, Edinburgh
  - NHS Greater Glasgow and Clyde/University of Glasgow, Glasgow
  - Ixworth GP Practice, Ixworth
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts and the London School of Medicine and Dentistry, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospital NHS Trust, Norwich

REFERENCES:
- [Derived] MacDonald TM, Williams B, Webb DJ, Morant S, Caulfield M, Cruickshank JK, Ford I, Sever P, Mackenzie IS, Padmanabhan S, McCann GP, Salsbury J, McInnes G, Brown MJ; British Hypertension Society Programme of Prevention And Treatment of Hypertension With Algorithm-based Therapy (PATHWAY). Combination Therapy Is Superior to Sequential Monotherapy for the Initial Treatment of Hypertension: A Double-Blind Randomized Controlled Trial. J Am Heart Assoc. 2017 Nov 18;6(11):e006986. doi: 10.1161/JAHA.117.006986. PMID 29151036